CLINICAL TRIAL: NCT00750360
Title: Study to Monitor the Safety and Reactogenicity of GlaxoSmithKline Biologicals' Influenza Split Vaccine FLUARIX™ Administered According to the Prescribing Information in Korean Subjects Aged More Than 6 Months of Age at the Time of Vaccination
Brief Title: Study to Monitor the Safety and Reactogenicity of Fluarix™ in Korean Subjects Aged > 6 Months of Age.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 218352/054
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Influenza; Korea; FluarixTM
MeSH Terms: conditions — Influenza, Human

ARMS (6):
- Unprimed, > 6 to < 72 Months (Experimental): Subjects aged > 6 months to < 72 months who were previously not vaccinated against influenza (unprimed).
  Interventions: Biological: FluarixTM
- Unprimed, ≥ 72 to < 108 Months (Experimental): Subjects aged ≥ 72 months to < 108 months who were previously not vaccinated against influenza (unprimed).
  Interventions: Biological: FluarixTM
- Primed, > 6 to < 72 Months (Experimental): Subjects aged > 6 months to < 72 months who previously received a vaccination against influenza (primed).
  Interventions: Biological: FluarixTM
- Primed, ≥ 72 to < 108 Months (Experimental): Subjects aged ≥ 72 months to < 108 months who previously received a vaccination against influenza (primed).
  Interventions: Biological: FluarixTM
- Primed, ≥ 108 to < 216 Months (Experimental): Subjects aged ≥ 108 months to < 216 months who previously received a vaccination against influenza (primed).
  Interventions: Biological: FluarixTM
- Primed, ≥ 216 Months (Experimental): Subjects aged ≥ 216 months who previously received a vaccination against influenza (primed).
  Interventions: Biological: FluarixTM

INTERVENTIONS:
Biological: FluarixTM — All subjects will receive a single dose of FluarixTM. For children less than 9 years of age who have not previously been vaccinated against influenza, a second dose will be given after an interval of at least 4 weeks (Group B).

SUMMARY:
The present study collects data on safety and reactogenicity of the vaccine in the local target population (600 or more subjects) as per the requirement of Korean Food and Drugs Administration (KFDA).

ELIGIBILITY:
Inclusion Criteria:

* A male or female > 6 months of age at the time of the first vaccination.
* Subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Free of obvious health problems as established by medical history and clinical examination judged by the investigator before entering into the study.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after vaccination.

Exclusion Criteria:

* Clinical signs of acute febrile illness at the time of entry into the study.
* Any treatment with immunosuppressive drugs, including oral and parenteral corticosteroids.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or previous severe reaction to influenza virus vaccine.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 883 (Actual)
Dates: Start 2003-10-03; Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 218352/054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 218352/054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 218352/054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 218352/054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 218352/054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 218352/054 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unprimed, > 6 to < 72 Months | Unprimed, ≥ 72 to < 108 Months | Primed, > 6 to < 72 Months | Primed, ≥ 72 to < 108 Months | Primed, ≥ 108 to < 216 Months | Primed, ≥ 216 Months
Started | 294 (Seven subjects enrolled in this group were not vaccinated and as such not included as "STARTED".) | 1 (One subject enrolled in this group was not vaccinated and as such not included as "STARTED".) | 384 | 79 | 46 | 71
Completed | 294 | 1 | 384 | 79 | 46 | 71
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unprimed, > 6 to < 72 Months | Unprimed, ≥ 72 to < 108 Months | Primed, > 6 to < 72 Months | Primed, ≥ 72 to < 108 Months | Primed, ≥ 108 to < 216 Months | Primed, ≥ 216 Months | Total
Number analyzed (Participants) | 294 | 1 | 384 | 79 | 46 | 71 | 875
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.7 (10.60) | 85.0 (0) | 38.3 (18.80) | 86.4 (10.60) | 132.7 (22.00) | 454.5 (174.40) | 73.2 (128.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 1 | 178 | 41 | 27 | 56 | 445
  Male | 152 | 0 | 206 | 38 | 19 | 15 | 430

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Severe Unsolicited Adverse Events
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Severe unsolicited adverse events are defined as adverse events which prevent normal, everyday activities
Time Frame: During the 21-day follow-up period (Day 0 to Day 20) after vaccination
Measure: Number; unit: participants
Arm/Group | Unprimed, > 6 to < 72 Months | Unprimed, ≥ 72 to < 108 Months | Primed, > 6 to < 72 Months | Primed, ≥ 72 to < 108 Months | Primed, ≥ 108 to < 216 Months | Primed, ≥ 216 Months
Number analyzed (Participants) | 294 | 1 | 384 | 79 | 46 | 71
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Reporting Solicited Local and General Adverse Events in Subjects Aged Less Than 72 Months.
Description: Solicited local adverse events assessed include induration, pain, redness, and swelling. Solicited general adverse events assessed include fever, shivering, and sweating/diaphoresis.
Time Frame: During the 4-day follow up (Day 0 to 3) after vaccination.
Measure: Number; unit: participants
Groups:
- Group B (Unprimed), > 6 Months to < 72 Months: Subjects aged > 6 months to < 72 months who were previously not vaccinated against influenza (unprimed).
- Group A (Primed), > 6 Months to < 72 Months: Subjects aged > 6 months to < 72 months who previously received a vaccination against influenza (primed).
Arm/Group | Group B (Unprimed), > 6 Months to < 72 Months | Group A (Primed), > 6 Months to < 72 Months
Number analyzed (Participants) | 294 | 384
participants
  Induration | 3 | 22
  Pain | 3 | 58
  Redness | 3 | 40
  Swelling | 2 | 36
  Fever | 7 | 9
  Shivering | 0 | 3
  Sweating/diaphoresis | 1 | 2

3. Secondary Outcome: Number of Participants Reporting Solicited Local and General Adverse Events in Subjects Aged 72 Months and Older.
Description: Solicited local adverse events assessed include induration, pain, redness, and swelling. Solicited general adverse events assessed include fatigue, fever, shivering, malaise, myalgia, headache, and sweating/diaphoresis.
Time Frame: During the 4-day follow up (Day 0 to 3) after vaccination.
Measure: Number; unit: participants
Groups:
- Group B (Unprimed), ≥ 72 Months to < 108 Months: Subjects aged ≥ 72 months to < 108 months who were previously not vaccinated against influenza (unprimed).
- Group A (Primed), ≥ 72 Months to < 108 Months: Subjects aged ≥ 72 months to < 108 months who previously received a vaccination against influenza (primed).
- Group A (Primed), ≥ 108 Months to < 216 Months: Subjects aged ≥ 108 months to < 216 months who previously received a vaccination against influenza (primed).
- Group A (Primed), ≥ 216 Months: Subjects aged ≥ 216 months who previously received a vaccination against influenza (primed).
Arm/Group | Group B (Unprimed), ≥ 72 Months to < 108 Months | Group A (Primed), ≥ 72 Months to < 108 Months | Group A (Primed), ≥ 108 Months to < 216 Months | Group A (Primed), ≥ 216 Months
Number analyzed (Participants) | 1 | 79 | 46 | 71
participants
  Pain | 0 | 23 | 7 | 10
  Redness | 0 | 11 | 7 | 4
  Swelling | 0 | 10 | 6 | 4
  Induration | 0 | 8 | 5 | 4
  Fatigue | 0 | 3 | 3 | 2
  Fever | 0 | 2 | 1 | 0
  Headache | 0 | 4 | 2 | 1
  Malaise | 0 | 1 | 1 | 1
  Myalgia | 0 | 6 | 3 | 5
  Shivering | 0 | 0 | 0 | 2
  Sweating/diaphoresis | 0 | 0 | 0 | 2

4. Secondary Outcome: Number of Participant Reporting Unsolicited Adverse Events.
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 21-day follow-up period (Day 0 to Day 20) after vaccination
Measure: Number; unit: participants
Arm/Group | Unprimed, > 6 to < 72 Months | Unprimed, ≥ 72 to < 108 Months | Primed, > 6 to < 72 Months | Primed, ≥ 72 to < 108 Months | Primed, ≥ 108 to < 216 Months | Primed, ≥ 216 Months
Number analyzed (Participants) | 294 | 1 | 384 | 79 | 46 | 71
participants | 28 | 0 | 67 | 12 | 6 | 3

5. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAE).
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Within 1 month following vaccination
Measure: Number; unit: participants
Arm/Group | Unprimed, > 6 to < 72 Months | Unprimed, ≥ 72 to < 108 Months | Primed, > 6 to < 72 Months | Primed, ≥ 72 to < 108 Months | Primed, ≥ 108 to < 216 Months | Primed, ≥ 216 Months
Number analyzed (Participants) | 294 | 1 | 384 | 79 | 46 | 71
participants | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Unprimed, > 6 to < 72 Months | Unprimed, ≥ 72 to < 108 Months | Primed, > 6 to < 72 Months | Primed, ≥ 72 to < 108 Months | Primed, ≥ 108 to < 216 Months | Primed, ≥ 216 Months
Serious Adverse Events (participants affected / at risk) | 1/294 | 0/1 | 0/384 | 0/79 | 0/46 | 0/71
Other Adverse Events (participants affected / at risk) | 9/294 | 0/1 | 90/384 | 27/79 | 10/46 | 11/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unprimed, > 6 to < 72 Months (N=294) | Unprimed, ≥ 72 to < 108 Months (N=1) | Primed, > 6 to < 72 Months (N=384) | Primed, ≥ 72 to < 108 Months (N=79) | Primed, ≥ 108 to < 216 Months (N=46) | Primed, ≥ 216 Months (N=71)
Kawasaki's disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Unprimed, > 6 to < 72 Months (N=294) | Unprimed, ≥ 72 to < 108 Months (N=1) | Primed, > 6 to < 72 Months (N=384) | Primed, ≥ 72 to < 108 Months (N=79) | Primed, ≥ 108 to < 216 Months (N=46) | Primed, ≥ 216 Months (N=71)
Pain (General disorders) | 3 | 0 | 58 | 23 | 7 | 10
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 40 | 11 | 7 | 4
Swelling (General disorders) | 2 | 0 | 36 | 10 | 6 | 4
Induration (General disorders) | 3 | 0 | 22 | 8 | 5 | 4
Fatigue (General disorders) | 0 | 0 | 1 | 3 | 3 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 4 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 6 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.